CLINICAL TRIAL: NCT01442857
Title: The Axillary Region in a High Resolution MRI. Imaging Before and After Brachial Plexus Block
Brief Title: The Axillary Region in a High Resolution MRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trygve Kjelstrup, MD, Section manager, Diakonhjemmet Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S-04115A
Record Dates: First submitted 2011-09-23; First posted 2011-09-29 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: MRI Scanner Configuration
Keywords: Magnetic Resonance Imaging; Nerve Net; Brachial Plexus; Nerve block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Block technique (Experimental): Active Comparator: Arm 1: catheter injection 40 ml of LA through the catheter
  Active Comparator: Arm 2: catheter and transarterial injection 20 + 10 ml transarterial block and 10 ml through the catheter
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — High resolution MRI of the brachial plexus

SUMMARY:
The axillary region is regularly used for brachial plexus block. The technique may be guided by nerve stimulation, ultrasound or a combination of nerve stimulation and ultrasound. Magnetic resonance imaging (MRI) has been beneficial in presenting anatomy of interest for regional anesthesia and in demonstrating spread of local anesthetic (LA). An axillary MRI-study at our department supported the suggestion of multiple rather than a single injection technique. Using a 0.5 Tesla open MR scanner in that study, the investigators were not able to distinguish terminal nerves from equally sized vessels. Therefore the investigators could not definitely answer whether the LA reached the pertinent nerves. The investigators have recently performed an axillary block study with a 3.0 Tesla scanner. Now the terminal nerves were identified and for each patient the investigators could observe if the LA reached the nerves.

The aim of this study was to demonstrate the anatomy of the brachial plexus in the axillary region at different levels. The investigators present the best pictures of the nerves with and without LA injected. The images are demonstrated in the axial and coronal plane.

DETAILED DESCRIPTION:
For upper limb surgery, the brachial plexus can be blocked at the interscalene, supraclavicular, infraclavicular and axillary level as an alternative to general anesthesia. The axillary block requires more deposits to achieve a complete block. MRI investigations are of interest to better understand the block specific distribution of LA. With the new MRI Achieva 3.0T X-series (Philips Electronics, Eindhoven the Netherlands), with resolutions beyond 100μm using 2k imaging, we expected new information also compared with the earlier axillary MRI publication from our department. In that former study we used a single deposit technique in an open 0.5 Tesla scanner. We could not in that study recognize the terminal nerves or determine if the LA reached the axillary plexus.

MRI publications of the brachial plexus mostly study the shoulder region and few are describing the axillary region. We did not find any article describing the axillary brachial plexus using a 3.0 Tesla high resolution MRI.

Ultrasound visualizes the plexus nerves in the axilla and demonstrates dynamically the spread of LA. This usually occurs in 2-dimensional images where the initially observed LA fades after some minutes. MRI provides more easy 3 - dimensional images also in oblique planes compared with ultrasound.

This study was done in order to demonstrate the relevant anatomy in the volunteers and the spread of LA in patients. We also present the used protocols and MRI - stacks after having optimized the configuration of the 3.0 MRI scanner.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - 2.
* Anatomic volunteers or patients scheduled for hand surgery

Exclusion Criteria:

* Nerulogic disease or sequela

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pattern of local anaesthetic spread in axillary plexus block patients compared to MR images from volunteers without local anaesthesia injected. | 3 years
  The optimized configuration of the 3.0 Tesla MRI scanner demonstrated detailed images from the volunteers and the patients. The image difference between the two groups was visualized and described.
  The investigators examined 9 volunteers and 9 patients. The volunteers were tested with different protocols in the 3.0 Tesla MRI providing anatomic pictures. The patients had two different brachial plexus blocks. Subsequently they were scanned with MRI and finally tested clinically for block efficacy before operation.

CONTACTS AND LOCATIONS:
Overall Officials: Øivind ØK Klaastad, PhD, MD, Study Director — Oslo University Hospital
Locations (1):
- The Intervention Centre, Rikshospitalet, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Kjelstrup T, Courivaud F, Klaastad O, Breivik H, Hol PK. High-resolution MRI demonstrates detailed anatomy of the axillary brachial plexus. A pilot study. Acta Anaesthesiol Scand. 2012 Aug;56(7):914-9. doi: 10.1111/j.1399-6576.2012.02703.x. Epub 2012 May 9. PMID 22571443
- See also: Link to The Intervention Centre, Oslo University Hospital — http://www.ivs.no